CLINICAL TRIAL: NCT03407716
Title: Ginseng as an Intervention to Decrease Cancer-Related Fatigue in Post-Treatment Cancer Survivors: A Randomized Controlled Pilot Study
Brief Title: Ginseng in Decreasing Cancer-Related Fatigue After Treatment in Cancer Survivors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC16C2; NCI-2017-02494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC16C2 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-03

CONDITIONS: Cancer Survivor; Stage I Breast Cancer AJCC v7; Stage I Colon Cancer AJCC v6 and v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage II Colon Cancer AJCC v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIA Colon Cancer AJCC v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIB Colon Cancer AJCC v7; Stage IIC Colon Cancer AJCC v7; Stage III Breast Cancer AJCC v7; Stage III Colon Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIA Colon Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIB Colon Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IIIC Colon Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (North American ginseng extract AFX-2) (Experimental): Patients receive North American ginseng extract AFX-2 PO BID on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: American Ginseng; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- GROUP II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. At the end of course 2, patients may optionally crossover to Group I to receive ginseng for an additional 28 days.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: American Ginseng — Given PO
  Other Names: ginseng; Ginseng Root; Panax quinquifolius
  Arms: Group I (North American ginseng extract AFX-2)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: GROUP II (placebo)
Other: Questionnaire Administration — Correlative studies

SUMMARY:
This randomized pilot trial studies how well North American ginseng extract AFX-2 (ginseng) works in decreasing cancer-related fatigue after treatment in cancer survivors. Ginseng may decrease fatigue in people who were treated for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of ginseng on decreasing cancer-related fatigue (CRF) in post-treatment cancer survivors as measured by Multidimensional Fatigue Symptom Inventory MFSI-Short Form (SF) at 28 and 56 days compared to placebo-controlled group.

SECONDARY OBJECTIVES:

I. To assess the acceptability and feasibility of ginseng as therapy for CRF in posttreatment cancer survivors.

II. To evaluate toxicities and tolerability associated with 2,000 mg per day of North American ginseng extract AFX-2 (panax quinquefolius) when used for cancer-related fatigue.

III. To explore the impact of ginseng on secondary endpoints, various dimensions of fatigue as measured by the other subscales of the MFSI-SF, Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form, as well as the single measure of fatigue (captured on Fatigue Linear Analogue Scale).

IV. To determine clinically significant changes in fatigue scores per the various measures of fatigue using the global impression of change.

TERTIARY OBJECTIVES:

I. To explore the relationship between ginseng therapy, inflammation biomarker adiponectin, and post-treatment cancer survivors? fatigue.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive North American ginseng extract AFX-2 orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo PO BID on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. At the end of course 2, patients may optionally crossover to Group I to receive ginseng for an additional 28 days.

After completion of study, patients are followed up at day 28 and 56.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proven breast cancer or colon cancer (stage I, II or III)
* Treated with chemotherapy and surgery
* Treatment has been completed (except hormone therapy) for >= 90 days prior to registration
* No known evidence of disease
* Men or women with a history of CRF as defined by a score >= 4 on the numeric analogue scale (0 ? 10) (Eligibility Question Fatigue Scale)
* Presence of CRF >= 30 days prior to registration
* Hemoglobin >= 11.0 g/dL obtained =< 180 days prior to registration
* Serum glutamic-oxaloacetic transaminase (SGOT) =< 1.5 x upper limit of normal (ULN) obtained =< 180 days prior to registration
* Creatinine =< 1.2 X ULN obtained =< 180 days prior to registration
* Ability to complete questionnaire(s) in English by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up of the study and optional crossover (if applicable)
* Willing to provide blood samples for correlative research purposes
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* CROSSOVER RE-REGISTRATION - INCLUSION CRITERIA
* Treatment cannot begin prior to re-registering to the crossover phase and will ideally begin =< 7 days after registration for the crossover phase

Exclusion Criteria:

* Hypersensitivity to ginseng
* Use of ginseng capsules for fatigue, within the last 12 months
* Uncontrolled hypertension >= 2 times as noted in medical history (diastolic blood pressure > 100, systolic > 160) =< 90 days prior to registration
* Currently using any other pharmacologic agent to specifically treat fatigue including psychostimulants, antidepressants, etc., although antidepressants used to treat items other than fatigue (such as hot flashes) are allowed if the patient has been on a stable dose for >= 30 days prior to registration and plans to continue for >= 30 days after registration; erythropoietin agents to treat anemia are allowed
* Known brain metastasis or primary central nervous system (CNS) malignancy
* Chronic oral or intravenous systemic steroid use (defined as being used on a regular basis or who have a problem that has required ongoing use of steroids in the last 180 days for greater than 7 days)
* Diabetes (defined by being on oral hypoglycemics or insulin)
* Psychiatric disorder such as severe depression, manic depressive disorder, obsessive compulsive disorder or schizophrenia; (defined per medical history)
* Major surgery =< 28 days prior to registration
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Treatable causes of fatigue have not been ruled out, at least by history and exam criteria, by the treating provider, such as uncontrolled pain, hypothyroidism, or insomnia; NOTE: if these are considered to be the primary cause for the patient?s fatigue then the patient is not eligible for this trial
* Patients with pain requiring opioid pain medication; NOTE: over the counter analgesics such as Tylenol or ibuprofen are allowed
* New use of Ambien and/or other benzodiazepines =< 30 days prior to registration
* New use of sleep aids including melatonin =< 30 days prior to registration
* Use of full anticoagulant doses of coumadin or heparin (exception: 1 mg/day of coumadin for preventing catheter clots is allowed)
* Use of monoamine oxidase inhibitors (MAOI) inhibitors
* Patients scoring greater than 4 on a 0 to 10 scale with regard to sleep troubles or pain
* Patients planning to start any type of cancer therapy during the 8 week, double blind, course of the study, once randomized on the study
* Patients with malnutrition, active infection, significant pulmonary disease and cardiovascular disease as determined by the physician as they could impact fatigue
* Use of any over the counter herbal/dietary supplement marketed for fatigue or energy (for example, products containing any type of ginseng, Rhodiola rosea, high doses of caffeine, guarana, or anything called an ?adaptogen?)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 180 days prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Change in general subscale of the Multidimensional Fatigue Symptom Inventory- Short Form (MFSI-SF) | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter

SECONDARY OUTCOMES:
Change in MFSI-SF emotional subscale | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter
Change in MFSI-SF general subscale | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter
Change in MFSI-SF mental subscale | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter
Change in MFSI-SF physical subscale | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter
Change in MFSI-SF vigor subscale | Baseline up to day 56
  Will be evaluated by taking the change from baseline in the general subscale of the MFSI-SF and comparing the two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used. Graphical procedures will include stream plots of individual patient scores and plots of average values over time for each treatment group. Supplemental tests on endpoints (paired t-test for continuous/ordinal data; McNemar?s test for binary data; and Bowker?s test for categorical data) will be utilized to deter
Change in the single item numeric analogue fatigue question | Baseline up to day 56
  Analysis will involve a t-test and Wilcoxon rank sum procedures (as appropriate).
Fatigue as measured by the National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) score | At day 28
  Analysis will involve a t-test and Wilcoxon rank sum procedures (as appropriate).
Fatigue as measured by the NIH PROMIS score | At day 56
  Analysis will involve a t-test and Wilcoxon rank sum procedures (as appropriate).
Incidence of adverse events as reported by the patient in a Ginseng Symptom Experience Diary | Up to day 56
  Any other possible side effects are recorded in the diary and assessed through nurse phone calls using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Descriptive statistics of frequency (percentage) will be used to summarize adverse event (AE) incidence and severity as measured by the CTCAE version 4.0 for each randomized arm separately. Toxicity data and other incidence rate-based endpoints will be compared across treatment groups using chi-square testing. Binomial confidence intervals for toxicity incidence rates will be constructed for each treatment group. The Gins
Perceived treatment efficacy as measured by the Subject Global Impression of Change | At 4 weeks
  Analysis will involve a t-test and Wilcoxon rank sum procedures (as appropriate). Descriptive statistics will be used to summarize the Global Impression of Change.
Perceived treatment efficacy as measured by the Subject Global Impression of Change | At 8 weeks
  Analysis will involve a t-test and Wilcoxon rank sum procedures (as appropriate). Descriptive statistics will be used to summarize the Global Impression of Change.

OTHER OUTCOMES:
Change in inflammation biomarkers (adiponectin, cortisol, IL-6) | Baseline up to day 84
  Cytokine levels and cortisol slopes will be described for the sample as a whole at baseline and at 28 days using means and frequencies. Relationships using Spearman correlation will be performed on fatigue measures, mood, and cytokine levels and cortisol slopes as well as evening cortisol levels at baseline. Baseline fatigue scores on the linear analogue scale will then be grouped into a dichotomous variable, (4 to 7 versus 8 to 10) to evaluate whether differences in cortisol and cytokine expression exist based on fatigue severity, using chi square analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Arring, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials